CLINICAL TRIAL: NCT00951262
Title: Development and Evaluation of a Life Review Program for Advanced Cancer Patients in Fuzhou, China
Brief Title: Intervention Study on Life Review Among Advanced Cancer Patients in Fuzhou, China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Enid Kwong, School of Nursing, The Hong Kong Polytechinich University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSEARS20090205002
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2009-08

CONDITIONS: Advanced Cancer
Keywords: life review; quality of life; advanced cancer patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- life review (Experimental): a life review program includes 3-session life review and formulation of a life review book as a gift for advanced cancer patients.
  Interventions: Behavioral: a life review program
- controlled group (No Intervention): the subjects in the controlled group do not receive the life review program

INTERVENTIONS:
Behavioral: a life review program — The life review program includes reviewing a life and formalating a life booklet. Reviewing a life consists of three weekly sessions separately addressing illness experience, adulthood life and childhood and adolescence life. Each session lasts about 30 to 60mintues.A booklet with photos documented significant life events will be produced as a gift for the subjects. The edition, photos and contents fo the booklet are determined by the subjects.
  Other Names: evaluative reminence
  Arms: life review

SUMMARY:
This study aims to develop a life review program and test its effectiveness on a sample of patients with advanced cancer patients receiving palliative care at home in Fuzhou.

DETAILED DESCRIPTION:
A life review program is mainly developed based on Erickson's theory, Confucius's teaching on human development, and the empirical findings of the researcher's preliminary study and pre-pilot study. The program covers reviewing a life for advanced cancer patients and formulating a booklet for them. A randomized controlled trial will be adopted for evaluation of this program. Eligible patients will be randomly assigned to the experimental group and the control group. The subjects in the experimental group will receive a life review program for three weeks. The outcome measure is quality of life (QOL), including domains of physical discomfort, food-related concerns, health care concerns, support, negative emotions, sense of alienation, existential distress and value of life. Subjects' QOL will be assessed before commencement of the program (T0) and one day (T1) and three weeks (T2) after the completion of the program for all subjects in two groups. Perceptions of the program will be elicited within three days after the program for subjects in the experimental group.Descriptive statistics will be used to analyze patients' personal information, disease related information, functional performance and QOL of advanced cancer patients. Repeated measures ANOVA will be used to measure QOL differences in between-group, within-group and interaction effects. Content analysis will be used to analyze the qualitative data collected.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are newly admitted to the study hospice
2. Patients who are suffering from cancer with metastasis made by a physician
3. Patients who know their diagnosis, prognosis and therapy
4. Patients' functional performance (the score of KPS) at or more than 50%
5. Patients who are adults (≥18 years old)
6. Patients who have no cognitive and verbal communication impairments

Exclusion Criteria:

1. Patients with planned treatments, such as chemotherapy, radiotherapy or surgery
2. Patients with psychiatric disorders
3. Patients who live outside Fuzhou since the following-up home visit services are not extended to those areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-02; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
quality of life | three weeks and six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Enid Kwong, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- The Fujian Hospice, Fuzhou, Fujian, China